CLINICAL TRIAL: NCT04629885
Title: A Phase 2b, Double-blind, Randomized, Parallel, Placebo-Controlled Study to Evaluate the 12-week Efficacy of Vagitocin in Postmenopausal Women With Symptoms of Vulvovaginal Atrophy
Brief Title: Study to Evaluate Efficacy of Vagitocin in Postmenopausal Women With Vulvovaginal Atrophy Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PepTonic Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXYPEP202; 2016-000158-36 (EudraCT Number)
Record Dates: First submitted 2017-05-08; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Vulvovaginal Atrophy
MeSH Terms: interventions — Oxytocin; Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin 400 IU (Experimental): 1mL Oxytocin 400 IU vaginal gel once daily for 12 weeks
  Interventions: Drug: Oxytocin 400 IU vaginal gel
- Placebo (Placebo Comparator): 1mL Placebo vaginal gel once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin 400 IU vaginal gel
  Other Names: Vagitocin
  Arms: Oxytocin 400 IU
Drug: Placebo — Matching placebo gel with identical appearance to the test product, used as reference treatment.
  Other Names: Placebo (for Vagitocin)
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo controlled Phase 2b study, divided in 2 parts:

* The main part of the study investigates the efficacy and safety of the Investigational Medicinal Product (IMP), intravaginally administered in glass syringes, on postmenopausal women with vulvovaginal atrophy symptoms.
* The exploratory part of the study investigates the efficacy and safety of the IMP, intravaginally administered in a laminate tube, on postmenopausal women with vulvovaginal atrophy symptoms.

A comparison of plasma levels of oxytocin when the IMP is administered by 2 different applicators will be investigated in a sub-group of patients.

In the main part, 160 subjects are enrolled and randomized to 2 different groups; 80 subjects receiving IMP and 80 subjects receiving placebo, in glass syringes. In the exploratory part of the study, 40 patients will be enrolled and randomized to 2 different groups; 30 subjects receiving IMP and 10 patients receiving placebo, in laminate tubes.

The study is conducted at 3 sites in Sweden, and comprises 5 visits: screening visit (Visit 0), randomization visit (Visit 1; Day 0), treatment follow-up visit (Visit 2; Week 4), end of treatment visit (Visit 3; Week 12) and a telephone follow-up visit (Visit 4; Week 14). All patients self-administer the IMP once daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 40-65 years at the time of screening, who are willing to participate in the study as indicated by signing the informed consent.
* Postmenopausal women with at least 24 months of spontaneous amenorrhea, or women who have had surgical bilateral oophorectomy with or without hysterectomy at least 6 weeks ago.
* Have ≤ 5% superficial cells in vaginal smear cytology at screening.
* Have a vaginal pH > 5.0 at screening.
* Have one moderate to severe vulvovaginal atrophy symptom (vulvar/vaginal irritation and itching, vaginal dryness, dysuria, dyspareunia or presence of vaginal bleeding associated with vaginal sexual activity) that has been identified by the subject as being the most bothersome to her.
* Have a body mass index (BMI) ≤32 kg/m2.
* Be judged by the Principal Investigator or Sub-investigator as being in otherwise good health based on a pre-study medical evaluation performed within 21 days prior to the initial dose of study medication. The medical evaluation findings must include a) a normal or clinically non-significant finding at physical examination, b) a normal or clinically non-significant heart rate, c) a mean sitting systolic blood pressure ≤150 mmHg and diastolic blood pressure ≤90 mmHg at screening. Hypertensive subjects controlled with stable medications, who have a blood pressure ≤150 mmHg (systolic) and ≤ 90 (diastolic) mmHg are suitable for inclusion, d) a normal or clinically non-significant finding at gynaecological examination, e) a normal mammography (no masses or other diagnosed findings suspected of being malignant) that has been performed within 36 months prior to initial dose of study medication, f) a normal or clinically non-significant finding at clinical breast examination (no masses or other findings suspected of being malignant), g) an acceptable Papanicolaou ("Pap") smear for subjects with an intact uterus and cervix (no dysplastic or malignant cells), h) laboratory values within normal limits or with non-significant deviations from normal values.
* Have an endometrial thickness of <4 mm as determined by vaginal ultrasonography, in women with an intact uterus.
* Be willing to abstain from vaginal sexual activity and the use of vaginal douching within 24 hours prior to vaginal pH measurements at screening and at Visits 2 and 3.

Exclusion Criteria:

* Currently hospitalized.
* Have a history or ongoing cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychological, or musculoskeletal disease or disorder that is clinically significant in the opinion of the Principal Investigator or Sub-Investigator.
* Have had or have any known or suspected tumor disease that is clinically significant in the opinion of the Principal Investigator or Sub-Investigator.
* Have a history of endometrial hyperplasia or uterine/endometrial, breast or ovarian cancer.
* Have a history of undiagnosed vaginal bleeding.
* Have an ongoing urogenital infection in spite of treatment at the randomization visit.
* Any contraindication to oxytocin therapy and allergy to the use of oxytocin and any components of the investigational drugs.
* Have a history of drug and/or alcohol abuse within one year of start of study.
* Have used any prescription or over-the-counter medications including phytoestrogens, herbal medicinal products or hormonal intra-uterine device with known estrogenic effects within 12 weeks prior to the screening visit.
* Have used any type of vaginal lubricants and moisturizers within 24 hours prior to the screening visit.
* Have used estrogen alone or estrogen/progestin for any of the following time periods: a) vaginal hormonal products (rings, creams, gels, vaginal suppositories) within 12 weeks prior to the screening visit, b) transdermal estrogen alone or estrogen/progestin products including percutaneous estrogen gels for at least 12 weeks prior to the screening visit, c) oral estrogen and/or progestin therapy within 12 weeks prior to the screening visit, d) intrauterine progestin therapy within 12 weeks prior to the screening visit, e) progestin implants and estrogen alone injectable drug therapy within 12 weeks prior to the screening visit, f) estrogen pellet therapy or progestational injectable drug therapy within 6 months prior to the screening visit.
* Have any reason, which in the opinion of the Principal Investigator or Sub-Investigator would prevent the subject from safely participating in the study or complying with protocol requirements.
* Have participated in another clinical study within 90 days prior to screening, have received an investigational drug within three months prior to the initial dose of study medication, or be likely to participate in another clinical study or receive another investigational medication during the study.
* Have contraindication to any planned study procedure.
* Pregnancy.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
Change in severity of the most bothersome VVA symptom. | Baseline and after 12 weeks of treatment.
  Change in severity of the VVA symptom (vulvar/vaginal irritation and itching, dyspareunia, vaginal dryness, dysuria or the absence or presence of vaginal bleeding associated with vaginal sexual activity [yes/no]) that has been self-identified by the subject as being the most bothersome to her at baseline.

SECONDARY OUTCOMES:
Change in vaginal pH | Baseline and 12 weeks of treatment.
  Change in vaginal pH (decrease is positive).
Change in % superficial cells | Baseline and 12 weeks of treatment.
  Change in % superficial cells in vaginal smear (increase is positive).
Change in maturation value | Baseline and 12 weeks of treatment.
  Change in maturation value (MV) (increase is positive). Maturation value is calculated using the percentage of parabasal cells, intermediate cells, and superficial cells in vaginal smear.
Change in summary score for the vulvovaginal atrophy symptoms. | Baseline and 12 weeks of treatment.
  Change in summary score for the VVA symptoms vulvar/vaginal irritation and itching, dyspareunia, vaginal dryness and dysuria (decrease is positive).
Change in severity of the most bothersome VVA symptom. | Baseline and 4 weeks of treatment.
  Change in severity of the VVA symptom (vulvar/vaginal irritation and itching, dyspareunia, vaginal dryness, dysuria or the absence or presence of vaginal bleeding associated with vaginal sexual activity [yes/no]) that has been self-identified by the subject as being the most bothersome to her at baseline.
Change in % superficial cells | Baseline and 4 weeks of treatment.
  Change in % superficial cells in vaginal smear (increase is positive).
Change in vaginal pH | Baseline and 4 weeks of treatment.
  Change in vaginal pH (decrease is positive).
Change in % parabasal cells | Baseline and 4 and 12 weeks of treatment.
  Change in % parabasal cells (decrease is positive).
Change in maturation value | Baseline and 4 weeks of treatment.
  Change in maturation value (MV) (increase is positive). Maturation value is calculated using the percentage of parabasal cells, intermediate cells, and superficial cells in vaginal smear.
Change in severity of the most bothersome VVA symptom. | Baseline and 4 and 12 weeks of treatment.
  Change in severity of the VVA symptom (vulvar/vaginal irritation and itching, dyspareunia, vaginal dryness, dysuria or the absence or presence of vaginal bleeding associated with vaginal sexual activity [yes/no]) that has been self-identified by the subject as being the most bothersome to her at baseline.
Change in Quality of Life evaluation parameters. | Baseline and 12 weeks of treatment
  Change in Quality of Life evaluation parameters.
Change in body weight. | Baseline and 12 weeks of treatment
  Change in body weight.
Change over time of clinical safety data. | Baseline and up to 14 weeks after first dose.
  Change over time of clinical safety data (adverse events, vital signs, physical, gynecological and breast examination findings, laboratory tests, transvaginal ultrasound and pap smear).

OTHER OUTCOMES:
Plasma concentrations of oxytocin administered by two different applicators. | 30 minutes pre-dose, pre-dose (t=0), 15, 30, 60, 120 and 240 minutes post-dose.
  Oxytocin levels in plasma measured in 20 subjects treated with Oxytocin administered in glass syringe and in 16 subjects treated with Oxytocin administered in laminate tube.

CONTACTS AND LOCATIONS:
Overall Officials: Aino Fianu Jonasson, MD, Principal Investigator — Kvinnoforskningsenheten K59, Karolinska Universitetssjukhuset, Huddinge
Locations (3):
- Sweden (3):
  - Kvinnoforskningsenheten K59, Karolinska Universitetssjukhuset, Huddinge
  - Kvinnokliniken, Norrlands Universitetssjukhus, Umeå
  - Kvinnokliniken, Akademiska sjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: No